CLINICAL TRIAL: NCT00296829
Title: Immunogenicity of Two Dosages of Inactivated, Split-Virion Influenza Vaccine Given by an Alternate Route in the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GID16
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Orthomyxoviridae Infection; Influenza; Myxovirus Infection
Keywords: Influenza;; Orthomyxoviruses;; Inactivated Split-virion influenza vaccine;; Elderly.
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Inactivated, split-virion influenza vaccine

SUMMARY:
All marketed influenza vaccines are injected by the intramuscular route. This study will test whether an influenza vaccine is effective when injected by other route than into the muscle. In order to prove this, the amount of antibodies in the blood will be measured before and after vaccination. In addition, the safety of both influenza vaccines will be tested by evaluating all serious reactions occurring after vaccination. The vaccine injected in this study is similar to the sponsor's marketed intramuscular influenza vaccine (Vaxigrip).

Primary Objective:

To demonstrate and compare the immune response of two dosages of influenza vaccine administered by an alternate route to the intramuscular administration of the vaccine.

Secondary Objectives:

* To compare the immune response 21 days after vaccination between each investigational group versus intramuscular group for each influenza strain.
* To describe the safety profile after the vaccination in each study group
* To describe the compliance of the two dosages of the vaccine administered by the alternate route with the European Medicine Agency.

Observational Objectives:

* To describe the safety profile during the 21-day period following an intramuscular revaccination in each group and the possibility of any reaction at the first injection site.
* To describe the pain at the injection site with a Visual Analog Scale and the acceptability of the injection using a questionnaire in each group.
* To describe the leakage appearing at the injection site immediately after the alternate route injection and to explore the relationship with immunogenicity.
* To evaluate the cellular mediated immune response in a subset of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 85 years on the day of inclusion
* Informed consent form signed
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Systemic hypersensitivity to egg proteins, chick proteins, or any of the vaccine components, in particular, neomycin, formaldehyde, and octoxinol 9, or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Febrile illness (oral temperature >= 37.5°C equivalent rectal temperature >= 38.0°C) on the day of inclusion
* Any vaccination or participation in another clinical trial in the four weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding six months, or long-term systemic corticosteroids therapy
* Chronic illness at a stage that could interfere with trial conduct or completion
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Blood or blood-derived products received in the past three months
* Vaccination planned in the four weeks following the first trial vaccination
* Previous vaccination against influenza (in the previous six months) with the trial vaccine or another vaccine
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1080
Dates: Start 2006-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (9):
- Australia (6):
  - Adelaide
  - Carina Heights
  - Inala
  - Kippa-Ring
  - Victoria
  - Westmead
- New Zealand (3):
  - Auckland
  - Dunedin
  - Hamilton

REFERENCES:
- [Derived] Holland D, Booy R, De Looze F, Eizenberg P, McDonald J, Karrasch J, McKeirnan M, Salem H, Mills G, Reid J, Weber F, Saville M. Intradermal influenza vaccine administered using a new microinjection system produces superior immunogenicity in elderly adults: a randomized controlled trial. J Infect Dis. 2008 Sep 1;198(5):650-8. doi: 10.1086/590434. PMID 18652550
- See also: Related Info — http://www.sanofipasteur.com